CLINICAL TRIAL: NCT03352817
Title: Study of Sexual Dysfunction and Place of Sexuality in Patients Included in a Cardiac Rehabilitation Program in Champagne-Ardenne
Brief Title: Study of Sexual Dysfunction in Patients Included in a Cardiac Rehabilitation Program in Champagne-Ardenne
Acronym: SexualDysf
Status: Completed | Type: Observational
Sponsor: CHU de Reims (Other)
Responsible Party: Sponsor
Other Study IDs: PZ17040
Record Dates: First submitted 2017-11-17; First posted 2017-11-24 (Actual); Last update posted 2018-05-18 (Actual); Status verified 2018-05

CONDITIONS: Patients With Heart Disease
MeSH Terms: interventions — Cardiac Rehabilitation

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients in cardiac rehabilitation: Eligible patients must have reached the age of majority, participate in a CR program at one of the centers cited, and agreed to respond to the study questionnaire voluntarily
  Interventions: Other: Cardiac rehabilitation

INTERVENTIONS:
Other: Cardiac rehabilitation — A questionnaire and an information sheet are provided. The questionnaire had to be completed anonymously and individually by the patient, to avoid any influence.

SUMMARY:
Sexual health is an important marker of individual quality of life and well-being of patients. Sexual dysfunction (SD) is common in patients with heart disease. Screening and management are recommended. Cardiac rehabilitation (CR) seems to be a privileged moment to address this problem, but the management is often insufficient. The main objective of the study was to evaluate the prevalence of SD in patients in CR in the Champagne-Ardenne region. Secondary objectives were to describe SD most frequently encountered, to identify risk factors of SD, to compare the feelings of patients about their sex life, before and after an acute cardiac event and to collect an estimate of the need for care by a dedicated sexology workshop. The investigators conducted an observational multicenter prospective study for descriptive and analytical purposes after approval by the Institutional review board. An anonymous questionnaire was distributed from June 1 to September 1, 2017 in patients participating in a cardiac rehabilitation program in the various centers in the region.

DETAILED DESCRIPTION:
Sexual health is an important marker of individual quality of life and well-being of patients. Sexual dysfunction (SD) is common in patients with heart disease. Screening and management are recommended. Cardiac rehabilitation (CR) seems to be a privileged moment to address this problem, but the management is often insufficient. The main objective of the study was to evaluate the prevalence of SD in patients in CR in the Champagne-Ardenne region. Secondary objectives were to describe SD most frequently encountered, to identify risk factors of SD, to compare the feelings of patients about their sex life, before and after an acute cardiac event and to collect an estimate of the need for care by a dedicated sexology workshop.

This prospective multicentre study was carried out in the cardiac rehabilitation centers of Champagne-Ardenne (Reims, Ardennes and Troyes ) between 1 June and 1 September 2017 by anonymous self-questionnaire.

Eligible patients must have reached the age of majority, participate in a CR program at one of the centers cited, and agreed to respond to the study questionnaire voluntarily. Sexual inactivity and celibacy were not exclusionary criteria because prior sexual behavior did not predict future behavior and the need for counseling. Patients were informed about the objectives and conduct of the study by a health professional during their rehabilitation program or in follow-up consultations with the cardiologist. If the patient agreed to participate in the study, a questionnaire and an information sheet was provided. The questionnaire had to be completed anonymously and individually by the patient, to avoid any influence. It was then put back in an enclosed opaque envelope, in a closed urn left near the cloakroom of each center.

Data are described as mean (± standard deviation) for quantitative variables and as a percentage for categorical variables. The Student or Wilcoxon-Mann Whitney test were used for the quantitative variables and chi-square or Fisher's exact test for categorical variables. The multivariate analysis of SD risk factors was performed by logistic regression. The Odds Ratio (OR) is reported with its 95% confidence interval (CI). The tests were bilateral with a threshold of significance at p <0.05.

ELIGIBILITY:
Inclusion Criteria:

* patients must have reached the age of majority, participate in a CR program at one of the centers cited, and agreed to respond to the study questionnaire voluntarily

Exclusion Criteria:

* <18yo

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Eligible patients must have reached the age of majority, participate in a CR program at one of the centers cited, and agreed to respond to the study questionnaire voluntarily
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2017-09-01 (Actual); Study Completion 2017-09-01 (Actual)

PRIMARY OUTCOMES:
Prevalence of sexual dysfunction in cardiac rehabilitation | Day 0
  Specific key measurements or observations used to measure the effect of experimental variables in a study, or for observational studies, to describe patterns of diseases or traits or associations with exposures, risk factors or treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Reims, Reims, France

IPD SHARING:
Plan to Share IPD: Undecided